CLINICAL TRIAL: NCT03603899
Title: Imaging and Understanding Bronchiolitis Obliterans Syndrome (BOS) in Lung Transplantation With Hyperpolarized 129Xenon MR Lung Imaging
Brief Title: Hp129 Xenon Imaging and BOS in Lung Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-4120
Record Dates: First submitted 2017-10-04; First posted 2018-07-27 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2024-09

CONDITIONS: Bronchiolitis Obliterans
MeSH Terms: conditions — Bronchiolitis Obliterans

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hp 129Xenon (Experimental): Participants will inhale up to 4 doses of Hp129Xenon; each dose will be no more than 1 liter.
  Interventions: Drug: Hp 129Xenon

INTERVENTIONS:
Drug: Hp 129Xenon — 129 Xenon is a noble gas with no taste or smell. It will be made slightly magnetic (also called hyperpolarizing) and then inhaled into the lungs to provide better pictures of the lungs during MRI.

SUMMARY:
The research is being conducted to develop new imaging methods that are sufficiently sensitive to allow for early diagnosis of BOS, a chronic allograft rejection affecting 50-60% of lung transplanted recipients who survive 5 years after transplant. Although lung transplantation has evolved into an effective therapeutic option for a large number of pediatric patients with end-stage pulmonary disease, long-term survival after lung transplantation is far worse than after the transplantation of other solid organs. This research may improve patient outcomes through earlier diagnosis of changes leading to BOS by obtaining image guided research biopsies of transplanted lung. Biopsies may be used for future research of ex vivo biomarkers of BOS and in the development of treatments through future clinical trials.

DETAILED DESCRIPTION:
This protocol aims to

* Develop new imaging methods that are sufficiently sensitive to allow early diagnosis of BOS.
* Improve patient treatment outcomes through earlier diagnosis of changes leading to BOS by obtaining image guided biopsies of transplanted lung.
* Provide image guided biopsies for use in future research of ex vivo biomarkers of BOS and in the development of treatments through future clinical trials.

The study will achieve these aims through a prospective, non-randomized, longitudinal, observational study that will recruit about 5 subjects a year for 5 years. The study will follow these post lung transplant patients at 6 months and 1 year with 129Xe MRI (Hyperpolarized 129Xenon Magnetic Resonance Imaging) and image guided bronchial biopsies to detect early BOS and to better understand BO disease progression. The biopsies will provide future research for rapid determination of cellular and molecular mechanisms that lead to BOS and to facilitate identification and validation of translatable pharmaceutical targets.

ELIGIBILITY:
Inclusion Criteria:

* Lung Transplantation within the last 10 years or being assessed for possible lung transplantation.
* Participant must be able to hold their breath for up to 16 seconds.

Exclusion Criteria:

* Standard MRI exclusion criteria
* Bleeding disorders
* Participant is claustrophobic or otherwise unable to tolerate the imaging
* Pregnancy or positive pregnancy test
* Symptoms of respiratory infection within the past two weeks.
* Baseline oximetry at MRI visit of less than 95% on room air or less than 95% on a previously prescribed dosage of oxygen delivered by nasal cannula.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Capture 129Xe and proton MRI Images for clinician assessment | 6 months post transplant
  Capture HP 129Xe and 1H MR images for clinician review for regional ventilation defects in post-transplant BOS patients during routine clinical visits

SECONDARY OUTCOMES:
Capture 129Xe and proton MRI Images for clinician assessment | 12 months post transplant
  Capture HP 129Xe and 1H MR images for clinician review for regional ventilation defects in post-transplant BOS patients during routine clinical visits

CONTACTS AND LOCATIONS:
Overall Officials: Jason Woods, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

DOCUMENTS (1):
  • Study Protocol (2017-09-19): https://cdn.clinicaltrials.gov/large-docs/99/NCT03603899/Prot_001.pdf